CLINICAL TRIAL: NCT06318078
Title: A Research Study to Understand the Impact and Cost-effectiveness of a Digital Health Platform for iCCM in Uganda
Brief Title: Buikwe Electronic Community Health Information System Impact Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Malaria Consortium (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: UG2024001
Record Dates: First submitted 2024-01-23; First posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-01

CONDITIONS: Malaria; Diarrhea; Pneumonia
MeSH Terms: conditions — Malaria; Diarrhea; Pneumonia

STUDY DESIGN:
Intervention Model Description: Cluster Randomised Control Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): 570 children will be allocated to the intervention arm and children in this arm will be assessed using the eCHIS digital tool.
  Interventions: Other: eCHIS
- Control (No Intervention): 570 children will be allocated to the intervention arm and children in this arm will be assessed using the standard care and paper based tools.

INTERVENTIONS:
Other: eCHIS — The electronic Community health Information System (eCHIS) is a Government of Uganda owned application used by community health workers for quality health assessments and improved reporting. The eCHIS intervention allows for the registration of longitudinal profiles for client centered care as well as provides care guidance to aid decision making. For its users, the app has a task tab for schedule management and dashboards for performance help management and impact tracking by supervisors. This app is interoperable with national reporting tools such as DHIS2. The app has ten workflows including registration of households and new persons, death reporting, iCCM assessment, treatment and referral follow up, stock monitoring, data synchronization, pregnancy registration, ANC danger signs and follow up, family planning registration, and screening (tuberculosis, hypertension, sickle cell, tobacco use and net use).
  Arms: Intervention

SUMMARY:
The purpose of the study is to investigate the impact of the eCHIS intervention on key child health outcomes.

DETAILED DESCRIPTION:
Following national guidelines, 2 VHTs per village will be supported to provide the full eCHIS community health package. In total 856 VHTs in Buikwe district will have been trained and equipped with the national strategy and operational guidelines on eCHIS as well as the VHT full package (iCCM+ and VHT basic package (reproductive health, immunization, nutrition) guidelines. The VHTs will be equipped with mobile devices and iCCM supplies to start the management of community-based health among children aged five years within their respective communities. A cross-sectional cluster randomized controlled trial (cRCT) will be used to establish study outcomes in children under 5 years in the intervention and control areas using mixed methods (qualitative and quantitative) of data collection.

A total sample size of 1,140 children under five: 570 children under five, per arm, was scientifically determined for the study. During data collection, several quality control measures will be applied to ensure the data recorded reflect the facts, responses, observations, and events. A standard operating procedure (SOP) with roles and responsibilities of the data collectors will be prepared to ensure standardized methods for capturing data. After endline data collection, difference-in-differences (DID) analysis will be done to derive an estimate of the intervention effect on odds of the study outcomes.

Results will be disseminated through agreed peer-review publications and international conferences. Malaria Consortium Uganda will work with relevant stakeholders at the Ministry of Health and Medic Mobile to disseminate findings nationally and throughout the study district.

ELIGIBILITY:
Inclusion Criteria:

* · Children between 3-59 months,

  * Being resident in the study area,
  * Consent to participate in the study obtained,
  * Willingness and ability of the child's guardians to comply with the study protocol for the duration of the study including attending a designated health centre if their child has malaria symptoms during the data collection period.

Exclusion Criteria:

* Children aged below 3 months and above 59 months
* Children resident outside the study areas
* Those who have not consented to participate in the study

Ages: 3 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1140 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Out Patient Department attendance (due to malaria, pneumonia and diarrhoea) | Over 1 year
  Attendance measured through baseline and endline surveys
Hospitalisation (due to malaria, pneumonia and diarrhoea) | Over 1 year
  Attendance measured through baseline and endline surveys
malaria related mortality in the community and health facilities | Over 1 year
  Malaria related mortality measured through routine data

CONTACTS AND LOCATIONS:
Overall Officials: John Baptist Bwanika, Principal Investigator — Malaria Consortium
Locations (1):
- Buikwe, Buikwe, Uganda

IPD SHARING:
Plan to Share IPD: No